CLINICAL TRIAL: NCT06206460
Title: Follow-up Assessment of the Randomized Controlled Trial: Open-label Placebo Treatment of Women With Premenstrual Syndrome: A Randomized Controlled Trial
Brief Title: Follow-up Assessment of a Trial of Open-label Placebos for Women With Premenstrual Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-02187; ub24Frey
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome; Open-label Placebo; RCT follow up
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open Label Placebo with Treatment Rationale
  Interventions: Other: Online Assessment
- Open Label Placebo without Treatment Rationale
  Interventions: Other: Online Assessment

INTERVENTIONS:
Other: Online Assessment — Online Assessment which consists of:
  * Sociodemographic data (life changes, medical and gynaecological history)
  * German PMS symptom diary retrospectively for last menstrual cycle
  * Quality of Life Inventory (SF-12)
  * Expectancy of relief

SUMMARY:
With the proposed study, the investigators aim to evaluate the long-term efficacy of the open-label placebo (OLP) intervention in premenstrual syndrome (PMS) and to contribute to a broader understanding of how OLPs work. It is planned to survey participants of the intervention groups (OLP+ and OLP-) regarding symptom intensity and impairment due to PMS after the conclusion of our randomized controlled trial (RCT) and intervention provision. Additionally, it will be examined if there is a difference between the OLP group with and without a treatment rationale (OPL+ vs. OLP-) across time. More precisely, it will be investigated whether participants of the intervention groups with and without treatment rationale experience any long-term improvement.

ELIGIBILITY:
Inclusion Criteria:

* Participants are willing to participate in the follow-up study
* Participants have the ability to use an electronic device with internet access to complete the online follow-up survey
* Participants give Informed consent
* Participants have a regular menstruation (i.e., no menopause; pregnancy; cycle inhibiting medication etc.)

Exclusion Criteria:

* Pregnancy or breastfeeding (currently or within the last three months)
* A severe psychological or somatic disease, affecting premenstrual complaints (e.g., cancer of the uterus or fallopian tubes)
* Commencement of the menopause, sterilization, or (part) resection of the uterus or fallopian tubes
* Changes in body mass index (i.e., under 18 or above 30)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 95 women who participated in the intervention groups of the RCT OPEN-LABEL PLACEBO TREATMENT OF WOMEN WITH PREMENSTRUAL SYNDROME: A RANDOMIZED CONTROLLED TRIAL (OLPPMS_1, SNCTP000002809, NCT03547661) and completed study participation (OLP+: N=48 and OLP-: N=47).
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Symptom intensity of premenstrual syndrome | One time assessment at baseline (the start day 1-3 of the next menstrual cycle retrospectively for the last luteal phase)
  The items of the German PMS [Premenstrual Syndrome] Symptom diary will be used to measure symptom intensity retrospectively for the last luteal phase ( i.e., PMS phase). The scale consists of 27 items measured on a 6-point Likert scale. A decrease in scores indicates an improvement in symptom intensity. The minimum score is zero; the maximum 162.
Interference of premenstrual syndrome | One time assessment at baseline (the start day 1-3 of the next menstrual cycle retrospectively for the last luteal phase)
  The items of the German PMS [Premenstrual Syndrome] Symptom diary will be used to measure interference retrospectively for the last luteal phase ( i.e., PMS phase).
  The scale consists of 3 items measured on a 6-point Likert scale. A decrease in scores indicates an improvement in interference. The minimum score is zero; the maximum 162.

SECONDARY OUTCOMES:
Quality of life (Short-Form-12) | One time assessment at baseline (the start day 1-3 of the next menstrual cycle retrospectively for the last luteal phase)
  Quality of life will be measured by means of the SF-12 (Short-Form-12) questionnaire retrospectively for the last luteal phase (i.e., PMS phase). The questionnaire comprises 12 questions, and quality of life is measured on a 6-point Likert scale. Two summary scores can be calculated: a mental component and a physical component score. Scores range from 0-100, with higher scores indicating better functioning.
Partnership satisfaction (Zufriedenheit in der Partnerschaft: ZIP) | One time assessment at baseline (the start day 1-3 of the next menstrual cycle retrospectively for the last luteal phase)
  Partnership satisfaction will be measured by means of the ZIP (Zufriedenheit in der Partnerschaft) questionnaire retrospectively for the last luteal phase (i.e., PMS phase). The questionnaire comprises 7 questions, and partnership satisfaction is measured on a 5-point rating scale. Scores range from 7 to 35.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel, Faculty of Psychology, Division of Clinical Psychology and Psychotherapy, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided